CLINICAL TRIAL: NCT02587533
Title: Peripheral Chemoreflex/Arterial Baroreflex Interaction in Patients With Electrical Carotid Sinus Stimulation
Acronym: ChemoBar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Charite University, Berlin, Germany (Other); Vanderbilt University School of Medicine (Other); Mayo Clinic (Other); University of Bristol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CRC-KliPha-004
Record Dates: First submitted 2015-10-13; First posted 2015-10-27 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Hypertension, Resistant to Conventional Therapy
Keywords: Baroreflex; Chemoreflex; Autonomic nervous system; Sympathetic activity; Muscle sympathetic nerve activity (MSNA); Microneurography; Electrical baroreflex stimulation; Resistant hypertension; Device-based therapy
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy | interventions — Dopamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Hypoxia without dopamine (Active Comparator): Target hemoglobin oxygen saturation (SpO2) 80%. No pharmacologic suppression of chemoreflex afferents. Readout: Responses to electrical baroreflex stimulation.
  Interventions: Other: Hypoxia without dopamine
- Hypoxia with dopamine (Active Comparator): Target hemoglobin oxygen saturation (SpO2) 80%. Counteracting pharmacologic suppression of chemoreflex afferents. Readout: Responses to electrical baroreflex stimulation.
  Interventions: Other: Hypoxia with dopamine
- Hyperoxia without dopamine (Active Comparator): Nearly complete hemoglobin oxygen saturation. No additional pharmacologic suppression of chemoreflex afferents. Readout: Responses to electrical baroreflex stimulation.
  Interventions: Other: Hyperoxia without dopamine
- Hyperoxia with dopamine (Active Comparator): Nearly complete hemoglobin oxygen saturation. Additional pharmacologic suppression of chemoreflex afferents. Readout: Responses to electrical baroreflex stimulation.
  Interventions: Other: Hyperoxia with dopamine

INTERVENTIONS:
Other: Hypoxia without dopamine — Target hemoglobin oxygen saturation (SpO2) 80%.
  Arms: Hypoxia without dopamine
Other: Hypoxia with dopamine — Target hemoglobin oxygen saturation (SpO2) 80%. Dopamine dose 3 µg/kg/min.
  Arms: Hypoxia with dopamine
Other: Hyperoxia without dopamine — Nearly complete hemoglobin oxygen saturation.
  Arms: Hyperoxia without dopamine
Other: Hyperoxia with dopamine — Nearly complete hemoglobin oxygen saturation. Dopamine dose 3 µg/kg/min.
  Arms: Hyperoxia with dopamine

SUMMARY:
Peripheral chemoreceptors and baroreceptors are located in close proximity in the carotid artery wall at the level of the carotid bifurcation. Baroreceptor stimulation lowers sympathetic activity and blood pressure. In contrast, chemoreceptor stimulation raises sympathetic activity and blood pressure. Thus, beneficial effects of electrical carotid sinus stimulation on blood pressure could be diminished by chemoreceptor overactivity and/or concomitant chemoreceptor activation through the device. Therefore, our study will assess baroreflex/chemoreflex interactions in patients with resistant hypertension equipped with carotid sinus stimulators. The study will inform us of potential additional anti-hypertensive benefits of simultaneous chemoreceptor denervation during electrode placement. Furthermore, the results may provide information about suitable electrode design to spare co-activation of peripheral chemoreceptors. Taken together, the study will help develop strategies for improving responder rate and efficacy of carotid sinus stimulators in patients with resistant hypertension.

DETAILED DESCRIPTION:
Patients with implanted devices for electrical baroreflex stimulation are recruited according to inclusion and exclusion criteria until good quality recordings have been obtained in 10 out of maximally 15 patients. After obtaining written informed consent patients will be investigated in the laboratory on one day. In up to 20% of the patients we may fail to find an appropriate nerve recording position. In these cases we will ask the patient to repeat the experiment.

Patients will be investigated in the post-absorptive state after emptying their bladder. During instrumentation and measurements they will rest in supine position. We will fix chest electrodes for ECG and impedance cardiography. A peripheral venous catheter will be introduced for later dopamine infusion. Cuffs will be used at the upper arm and the finger in order to monitor blood pressure and to allow for pulse-contour analysis. Finally, we will search for a suitable nerve recording position in the peroneal nerve for recordings of muscle sympathetic nerve activity (MSNA, postganglionic vasoconstrictor sympathetic drive). All bioelectric signals will be recorded continuously for the duration of the experiments.

After the preparations baseline recordings will be performed. Subsequently, the electrical baroreflex stimulator is switched OFF and ON repeatedly (toggling) under normoxic conditions. Every OFF and ON state will last for 4 minutes. Oscillometric blood-pressure readings are taken every two minutes so as to acquire two readings per stimulation period. Toggling under normoxia is meant to ensure that the patient is a responder at the experimental day and to rule out that the blood pressure rises are too high off stimulation (safety concern). Afterwards, the breathing gas will be changed in order to have the patient inhale a hypoxic or hyperoxic mixture in a blinded manner. After reaching a stable ventilatory and autonomic state, stimulator toggling and blood-pressure measurements will be repeated. The same procedures will take place after establishing the opposite oxygenation state. Stimulation will be ON in between the oxygen states implying that the first switches will be OFF switches with all oxygenation conditions. Afterwards, the last oxygenation state will be maintained and additional low-dose dopamine infusion will be applied. Again, the electrical baroreflex stimulator will be switched off and on repeatedly and blood-pressure readings are taken. During the last two stimulator toggling states of each oxygenation level, venous blood samples are drawn for hormone measurements and inert gas rebreathing will take place for cardiac output determination. Finally, the correct positioning of the microneurography electrode is checked again.

The duration of such an experiment depends on the time needed to find the sympathetic nerve bundles before the measurements and during the experiment, in case the recording position gets lost. However, experiments will rarely exceed 5 hours in total.

ELIGIBILITY:
Inclusion Criteria:

* Implanted device for electrical baroreflex stimulation.
* The patient is a 'responder', i. e. carotid-sinus stimulation causes a drop in systolic arterial pressure by at least 15 mmHg.
* The patient gave informed consent.

Exclusion Criteria:

* The patient is an investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
* The mental condition renders the patient unable to understand the nature, scope, and possible consequences of the study.
* The patient is unlikely to comply with the protocol.
* The patient is pregnant or breast-feeding.
* Hypoxic conditions for half an hour are considered harmful, e. g. in patients with shunts.
* History of drug or alcohol abuse.
* Discontinuation of diuretic medication for one day is considered harmful. (Reason: Bladder distension is a sympathoexcitatory stimulus and shortens experimental time. In order to prevent these shortcomings three measures are taken: Dispensation with beverages and diuretics as well as complete bladder voiding immediately before the experiment.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity (MSNA) | Over 24 minutes of stable de/oxygenation +/- dopamine infusion.
  Muscle sympathetic nerve activity (MSNA) will be determined as burst frequency, i. e. as the number of bursts per minute [bursts/min]. In responders, electrical carotid sinus stimulation will lead to a decline in MSNA: [-]MSNA. According to our primary hypothesis, [-]MSNA during hyperoxic conditions ([-]MSNA_hyperoxia) is larger than during hypoxia ([-]MSNA_hypoxia). Therefore, the primary endpoint of the study is the difference [-]MSNA_hyperoxia - [-]MSNA_hypoxia. The study is successful as soon as the difference between the reduction in the hyperoxic and the hypoxic condition is significantly different from zero. A positive value would confirm our primary hypothesis. In case of a negative difference, we would conclude that the potency of electrical baroreflex stimulation to lower sympathetic activity is larger under conditions of an activated chemoreflex.

SECONDARY OUTCOMES:
Systolic blood pressure (SBP) | Over 24 minutes of stable de/oxygenation +/- dopamine infusion.
  In responders, electrical carotid sinus stimulation will lead to a decline in systolic blood pressure: [-]SBP. According to our primary hypothesis, [-]SBP during hyperoxic conditions ([-]SBP_hyperoxia) is larger than during hypoxia ([-]SBP_hypoxia). Therefore, the secondary endpoint of the study is the difference [-]SBP_hyperoxia - [-]SBP_hypoxia. A positive value would confirm our secondary hypothesis. If the difference turns out to be negative, we would conclude that the potency of electrical baroreflex stimulation to lower blood pressure is larger under conditions of an activated chemoreflex. However, such a finding would not necessarily imply that chemoreceptor activation is a prerequisite for optimal baroreflex activation therapy because SBP *level* could be lower with *inactive* chemoreceptors.

OTHER OUTCOMES:
End-tidal partial carbon dioxide pressure (etCO2) | Over 24 minutes of normoxia.
  Electrical carotid sinus stimulation may lead to co-activation of carotid body chemoreceptors which would result in increased ventilation and etCO2 reduction. According to our hypothesis, etCO2 is higher without than with electrical baroreflex stimulation. Hence, the endpoint is the difference etCO2,OFF - etCO2,ON.
  EtCO2 will be assessed during normoxia. Argument against hypoxia: The hypoxic challenge is expected to increase ventilation. The ensuing etCO2 drop would represent a confounder. Thus, we seek for normal etCO2 levels during hypoxia by adding variable tiny amounts of CO2 to the breathing gas. (Note: This is not an intervention but avoids an important confounder, namely etCO2 changes.) Argument against hyperoxia: Carotid body chemosensors may be desensitized to electrical stimulation during hyperoxia.
Individual responses (MSNA, BP) without dopamine | Over 24 minutes of stable de/oxygenation.
  MSNA and blood pressure responses to stimulation during normoxia and hyperoxia on an individual basis.
Individual responses (MSNA, BP) with dopamine | Over 24 minutes of dopamine infusion.
  Low-dose dopamine infusion is another means to simulate hyperoxic conditions. MSNA and blood pressure responses to stimulation with and without dopamine are to be compared.
MSNA burst incidence | Over 24 minutes of stable de/oxygenation +/- dopamine infusion.
  Changes in sympathetic activity measured as burst incidence (sympathetic bursts per 100 heart beats) and total activity (area under the sympathetic bursts).
Diastolic and mean blood pressure (DBP, MBP) | Over 24 minutes of stable de/oxygenation +/- dopamine infusion.
  Blood pressure responses to stimulation during normoxia, hyperoxia, and dopamine infusion.
Sympathetic and cardiac baroreflex sensitivity. | Over 24 minutes of stable de/oxygenation +/- dopamine infusion.
  Differences in the relationship between changes in sympathetic activity or heart interval and blood pressure.
Ventilation | Over 24 minutes of stable de/oxygenation +/- dopamine infusion.
  Air volume flow [L/min]

CONTACTS AND LOCATIONS:
Overall Officials: Jens Tank, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, LSX, Germany

REFERENCES:
- [Background] Grassi G. Counteracting the sympathetic nervous system in essential hypertension. Curr Opin Nephrol Hypertens. 2004 Sep;13(5):513-9. doi: 10.1097/00041552-200409000-00006. PMID 15300157
- [Background] Eckberg DL. Carotid baroreflex function in young men with borderline blood pressure elevation. Circulation. 1979 Apr;59(4):632-6. doi: 10.1161/01.cir.59.4.632. PMID 421303
- [Background] Somers VK, Mark AL, Abboud FM. Potentiation of sympathetic nerve responses to hypoxia in borderline hypertensive subjects. Hypertension. 1988 Jun;11(6 Pt 2):608-12. doi: 10.1161/01.hyp.11.6.608. PMID 3391673
- [Background] Trzebski A, Tafil M, Zoltowski M, Przybylski J. Increased sensitivity of the arterial chemoreceptor drive in young men with mild hypertension. Cardiovasc Res. 1982 Mar;16(3):163-72. doi: 10.1093/cvr/16.3.163. PMID 6805956
- [Background] McBryde FD, Abdala AP, Hendy EB, Pijacka W, Marvar P, Moraes DJ, Sobotka PA, Paton JF. The carotid body as a putative therapeutic target for the treatment of neurogenic hypertension. Nat Commun. 2013;4:2395. doi: 10.1038/ncomms3395. PMID 24002774
- [Background] Abdala AP, McBryde FD, Marina N, Hendy EB, Engelman ZJ, Fudim M, Sobotka PA, Gourine AV, Paton JF. Hypertension is critically dependent on the carotid body input in the spontaneously hypertensive rat. J Physiol. 2012 Sep 1;590(17):4269-77. doi: 10.1113/jphysiol.2012.237800. Epub 2012 Jun 11. PMID 22687617
- [Background] Sinski M, Lewandowski J, Przybylski J, Bidiuk J, Abramczyk P, Ciarka A, Gaciong Z. Tonic activity of carotid body chemoreceptors contributes to the increased sympathetic drive in essential hypertension. Hypertens Res. 2012 May;35(5):487-91. doi: 10.1038/hr.2011.209. Epub 2011 Dec 8. PMID 22158114
- [Background] Paton JF, Deuchars J, Li YW, Kasparov S. Properties of solitary tract neurones responding to peripheral arterial chemoreceptors. Neuroscience. 2001;105(1):231-48. doi: 10.1016/s0306-4522(01)00106-3. PMID 11483315
- [Background] Somers VK, Mark AL, Abboud FM. Interaction of baroreceptor and chemoreceptor reflex control of sympathetic nerve activity in normal humans. J Clin Invest. 1991 Jun;87(6):1953-7. doi: 10.1172/JCI115221. PMID 2040688
- [Background] Paton JF, Sobotka PA, Fudim M, Engelman ZJ, Hart EC, McBryde FD, Abdala AP, Marina N, Gourine AV, Lobo M, Patel N, Burchell A, Ratcliffe L, Nightingale A. The carotid body as a therapeutic target for the treatment of sympathetically mediated diseases. Hypertension. 2013 Jan;61(1):5-13. doi: 10.1161/HYPERTENSIONAHA.111.00064. Epub 2012 Nov 19. No abstract available. PMID 23172927
- [Background] Despas F, Lambert E, Vaccaro A, Labrunee M, Franchitto N, Lebrin M, Galinier M, Senard JM, Lambert G, Esler M, Pathak A. Peripheral chemoreflex activation contributes to sympathetic baroreflex impairment in chronic heart failure. J Hypertens. 2012 Apr;30(4):753-60. doi: 10.1097/HJH.0b013e328350136c. PMID 22241144
- [Background] Wennergren G, Little R, Oberg B. Studies on the central integration of excitatory chemoreceptor influences and inhibitory baroreceptor and cardiac receptor influences. Acta Physiol Scand. 1976 Jan;96(1):1-18. doi: 10.1111/j.1748-1716.1976.tb10166.x. PMID 1251739
- [Background] Heusser K, Tank J, Engeli S, Diedrich A, Menne J, Eckert S, Peters T, Sweep FC, Haller H, Pichlmaier AM, Luft FC, Jordan J. Carotid baroreceptor stimulation, sympathetic activity, baroreflex function, and blood pressure in hypertensive patients. Hypertension. 2010 Mar;55(3):619-26. doi: 10.1161/HYPERTENSIONAHA.109.140665. Epub 2010 Jan 25. PMID 20101001
- [Background] Schroeder C, Heusser K, Brinkmann J, Menne J, Oswald H, Haller H, Jordan J, Tank J, Luft FC. Truly refractory hypertension. Hypertension. 2013 Aug;62(2):231-5. doi: 10.1161/HYPERTENSIONAHA.113.01240. Epub 2013 May 20. No abstract available. PMID 23690343
- [Background] Jordan J, Heusser K, Brinkmann J, Tank J. Electrical carotid sinus stimulation in treatment resistant arterial hypertension. Auton Neurosci. 2012 Dec 24;172(1-2):31-6. doi: 10.1016/j.autneu.2012.10.009. Epub 2012 Nov 9. PMID 23146623
- [Background] Janssen C, Beloka S, Kayembe P, Deboeck G, Adamopoulos D, Naeije R, van de Borne P. Decreased ventilatory response to exercise by dopamine-induced inhibition of peripheral chemosensitivity. Respir Physiol Neurobiol. 2009 Sep 30;168(3):250-3. doi: 10.1016/j.resp.2009.07.010. Epub 2009 Jul 18. PMID 19619673
- [Background] Niewinski P, Tubek S, Banasiak W, Paton JF, Ponikowski P. Consequences of peripheral chemoreflex inhibition with low-dose dopamine in humans. J Physiol. 2014 Mar 15;592(6):1295-308. doi: 10.1113/jphysiol.2013.266858. Epub 2014 Jan 6. PMID 24396060
- [Background] Niewinski P, Janczak D, Rucinski A, Jazwiec P, Sobotka PA, Engelman ZJ, Fudim M, Tubek S, Jankowska EA, Banasiak W, Hart EC, Paton JF, Ponikowski P. Carotid body removal for treatment of chronic systolic heart failure. Int J Cardiol. 2013 Oct 3;168(3):2506-9. doi: 10.1016/j.ijcard.2013.03.011. Epub 2013 Mar 29. PMID 23541331
- [Background] Lipp A, Schmelzer JD, Low PA, Johnson BD, Benarroch EE. Ventilatory and cardiovascular responses to hypercapnia and hypoxia in multiple-system atrophy. Arch Neurol. 2010 Feb;67(2):211-6. doi: 10.1001/archneurol.2009.321. PMID 20142529
- [Background] Breskovic T, Valic Z, Lipp A, Heusser K, Ivancev V, Tank J, Dzamonja G, Jordan J, Shoemaker JK, Eterovic D, Dujic Z. Peripheral chemoreflex regulation of sympathetic vasomotor tone in apnea divers. Clin Auton Res. 2010 Apr;20(2):57-63. doi: 10.1007/s10286-009-0034-1. Epub 2009 Oct 10. PMID 19820987